CLINICAL TRIAL: NCT02012361
Title: Inspired Helium for Ischemic Protection During Knee Replacement Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201400033
Record Dates: First submitted 2013-12-10; First posted 2013-12-16 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Ischemia
Keywords: Ischemic preconditioning; Human limb ischemia; Total knee arthroplasty; Supplemental inspired helium
MeSH Terms: conditions — Ischemia | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): This group will be treated as any other patient would. Their anesthesia will be conducted as per routine with a target Fraction of inspired oxygen concentration (FiO2) of 0.25. During the course of the operation a small muscle biopsy will be collected.
  Interventions: Procedure: Control Group; Procedure: Muscle Biopsy
- Single-Dose Heliox Group (Active Comparator): This group will be treated with a single dose of inspired 75/25 heliox (75% helium 25% oxygen) breathed continuously for 15 minutes prior to the inflation of the surgical tourniquet. During the course of the operation a small muscle biopsy will be collected.
  Interventions: Procedure: Single-Dose Heliox Group; Procedure: Muscle Biopsy

INTERVENTIONS:
Procedure: Control Group — This group will be treated as any other patient would. Their anesthesia will be conducted as per routine with a target FiO2 of 0.25, (25%oxygen / 75%nitrogen) the only exception being that they will not be treated with inspired heliox.
  Arms: Control Group
Procedure: Single-Dose Heliox Group — This group will be treated with a single dose of inspired 75/25 heliox (75% helium 25% oxygen) breathed continuously for 15 minutes over any convenient window prior to the inflation of the surgical tourniquet. This will be the only change in their clinical care. Their anesthesia will be conducted as per routine and as the anesthesia team sees fit with a target FiO2 of 0.25, the only exception being that they will receive 75/25 heliox prior to the inflation of the tourniquet.
  Arms: Single-Dose Heliox Group
Procedure: Muscle Biopsy — During the course of the operation a small muscle biopsy will be collected.

SUMMARY:
The purpose of this study is to determine whether breathing in helium reduces indications of injury to the skeletal muscle seen in blood tests after knee replacement surgery.

The ability to reduce the risk of skeletal muscle injury may help improve patient safety by providing protection to the area of the body having its blood supply interrupted during a particular surgery.

DETAILED DESCRIPTION:
During hospitalization, beginning the day after surgery, additional tests will be added to the daily standard of care blood samples. When daily blood samples are not ordered as part of a study participants care after surgery, blood samples only for the study tests, may be done.

Up to 60 study participants will be selected to be in one of two possible groups.

After hospital discharge the study participants physical therapist will be contacted for copies of the notes and reports about the participants progress in physical therapy. This information will be used to evaluate if the different breathing gases have any impact on how quickly people recover after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an elective total knee arthroplasty
* > 18 years of age
* Expected to require inhaled oxygen concentrations < 25%
* Able to provide informed consent

Exclusion Criteria:

* Expected to require inhaled oxygen concentrations > 25%
* < 18 years of age
* Member of a defined vulnerable population (e.g. pregnant, mentally handicapped, prisoners, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Expression of serum markers | up to 5 days
  Post-operative expression of serum markers of injury to the skeletal muscle after knee arthroplasty.
  The primary endpoint will be detection of a decrease in the peak increase of CK detectable in the blood. A 15% decrease will be considered clinically significant.

SECONDARY OUTCOMES:
Recovery of quadriceps function | Up to one year
  Length of time of transition from a walker to a cane.

OTHER OUTCOMES:
Post-surgical time course of potassium | up to 5 days
  Changes in the time course of the peak level of expression of potassium will be analyzed.
Post-surgical time course of urea (BUN) | up to 5 days
  Changes in the time course of the peak level of expression of urea (BUN) will be analyzed.
Post-surgical time course of lactic acid | up to 5 days
  Changes in the time course of the peak level of expression of lactic acid will be analyzed.
Post-surgical time course of lactate dehydrogenase | up to 5 days
  Changes in the time course of the peak level of expression of lactate dehydrogenase will be analyzed..
Post-surgical time course of aldolase | up to 5 days
  Changes in the time course of the peak level of expression of aldolase will be analyzed.
Post-surgical time course of creatinine phosphokinase (CK) | up to 5 days
  Changes in the time course of the peak level of expression of creatinine phosphokinase (CK) will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron R. Smith, M.D., Ph.D., Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No